CLINICAL TRIAL: NCT06185517
Title: French Translation and Validation of the Michigan Retinal Degeneration Questionnaire and the Michigan Vision-Related Anxiety Questionnaire in a Cohort of People With Hereditary Retinal Degeneration.
Brief Title: Validation of Questionnaire in Retinal Degeneration
Acronym: VQDR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Collaborators: Street Lab (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P22-07
Record Dates: First submitted 2023-06-16; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-06

CONDITIONS: Retinal Degeneration
MeSH Terms: conditions — Retinal Degeneration

STUDY DESIGN:
Intervention Model Description: Comprehension phase:
  After an initial translation of the questionnaires into French, the aim of this of this phase is to ensure the level of understanding of each and potential suggestions, during a personal or telephone interview.
  Validation phase:
  The aim is to validate the French translation of the Michigan Retinal Degeneration Questionnaire (MRDQ) and the Michigan Vision-Related Anxiety Questionnaire (MVAQ), and in particular to assess: internal validity, construct validity, acceptability, reliability, sensitivity, specificity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehension Phase (Experimental): After an initial translation of the questionnaires into French, the aim of this phase is to ascertain the level of understanding of each questionnaire item and any suggestions, during a telephone or face-to-face interview.
  Interventions: Diagnostic Test: Questionnaire translation and validation
- Validation Phase (Experimental): The aim is to validate the French translation of the Michigan Retinal Degeneration Questionnaire (MRDQ) and the Michigan Vision-Related Anxiety Questionnaire (MVAQ).
  Interventions: Diagnostic Test: Questionnaire translation and validation

INTERVENTIONS:
Diagnostic Test: Questionnaire translation and validation — Michigan Retinal Degeneration Questionnaire (MRDQ) and the Michigan Vision-Related Anxiety Questionnaire (MVAQ). Validation of a French translation

SUMMARY:
While inherited retinal diseases are well characterized anatomically and functionally, it is also essential to understand their impact on patients' quality of life, from their ability to perform the tasks of daily living to the psychological impact of the disease on patients. Questionnaires (PRO, Patient-Reported Outcomes) are important tools for assessing this impact. However, PROs validated in French are rare, and often poorly adapted to populations with hereditary retinal degeneration. New PROs particularly adapted to retinal degeneration have recently been validated in English: the Michigan Retinal Degeneration Questionnaire (MRDQ) and the Michigan Vision-Related Anxiety Questionnaire (MVAQ). Validation of a French translation will provide a standardized, reliable tool for French-speaking patients, and enable these questionnaires to be used in gene therapy clinical trials, to assess the efficacy of treatments and their impact on patients' quality of life.

DETAILED DESCRIPTION:
Interventional research of category 2 with minimal risks and constraints. This is a prospective, monocentric, longitudinal, non-randomized study to validate the translation of questionnaires to assess abilities in daily living tasks and the potential psychological repercussions of visual impairment in various hereditary retinal dystrophies.

The research will be conducted in two distinct phases:

Comprehension phase and validation phase

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age: 18 to 80
* Sufficient knowledge of the French language to ensure understanding of the tasks to be performed and the instructions received.
* Signed consent after being informed by the investigator.
* Affiliation with health insurance.
* Affected by one of the following rare pathologies, with different levels of visual field, acuity and contrast sensitivity impairment:
* Non-syndromic rod-cone dystrophy (retinopathy pigmentosa, RP): diagnosis confirmed by a specialist.
* Non-syndromic rod-cone dystrophy: diagnosis confirmed by a specialist.
* Non-syndromic Stargardt's disease: diagnosis confirmed by a specialist.
* Non-syndromic congenital night blindness: diagnosis confirmed by a specialist.
* Non-syndromic achromatopsia: diagnosis confirmed by a specialist.

Exclusion Criteria:

* Pregnancy
* Inability to give informed consent.
* Cataract surgery within 3 months of inclusion.
* Hearing impairment that may interfere with comprehension during the interview.
* Functional amblyopia.
* Inability to comply with instructions to perform study tasks or study visits.
* Drug treatment that may cause motor, visual or cognitive impairment (PSAs, neuroleptics, etc.) or that may interfere with study assessments.
* Other uncontrolled ophthalmic conditions that may interfere with evaluation.
* Participation in another clinical trial that may interfere with the present study.
* Patient under guardianship, curatorship or legal protection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Reliability | 2 months
  will be assessed using intra-class correlations (ICC) between questionnaire measures in test-retest.
Acceptability | 2 months
  will be assessed by analyzing a comprehension questionnaire administered to participants.
Internal validity, | 2 months
  Internal validity is crucial to ensure that the questionnaire questions correctly measure the concept under study. It is assessed by examining the correlations between similar questions. High correlations indicate good internal validity, which means that the questionnaire is reliable and accurate for assessing the target concept.
Construct validity | 2 months
  Will be assessed by examining the relationships between questionnaire scores and other theoretically related measures. High correlations with similar measures and low correlations with unrelated measures indicate good construct validity.
Sensitivity | 2 months
  Will be assessed by analysing the questionnaire's ability to detect significant differences between groups of participants with different levels of disease severity. A sensitive questionnaire will make it possible to identify subtle differences between groups and will therefore be more useful for assessing the impact of the disease on patients' quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle AUDO, Principal Investigator — Centre Hospitalier National d'Ophtalmologie